CLINICAL TRIAL: NCT00719472
Title: A Phase III Multicenter, Open-label Study of Rituximab Alternative Dosing Rate in Patients With Previously Untreated Diffuse Large B-cell or Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of Rituximab Alternative Dosing Rate in Patients With Previously Untreated Diffuse Large B-cell or Follicular Non-Hodgkin's Lymphoma (RATE)
Acronym: RATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U4391g
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Results first posted 2012-06-26 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Follicular NHL; NHL; Large B-Cell NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; COP protocol 2; Analgesics; Antipyretics; Histamine Antagonists

ARMS (1):
- Rituximab 375 mg/m^2 (Experimental): Patients received 6 or 8 21-day cycles of CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone) or CVP (cyclophosphamide, vincristine, prednisone) in combination with rituximab 375 mg/m^2 administered by intravenous (IV) infusion on Day 1 of each cycle.
  Interventions: Drug: Rituximab; Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone); Drug: CVP (cyclophosphamide, vincristine, prednisone); Drug: Analgesic/antipyretic and antihistamine drugs

INTERVENTIONS:
Drug: Rituximab — During Cycle 1 rituximab was administered at an initial rate of 50 mg/hour. In the absence of infusion toxicity during Cycle 1, the infusion rate was escalated by 50 mg/h increments every 30 minutes to a maximum rate of 400 mg/hour. In case of infusion-related reactions, the infusion was interrupted or the infusion rate reduced. In case of Grade 3/4 infusion reactions, the rituximab infusion was discontinued and medical treatment provided. If the rituximab infusion in Cycle 1 was tolerated without a serious adverse event (AE) or Grade 3/4 infusion-related AE, as judged by the investigator, infusions in Cycle 2 onwards were administered as follows: 20% of the total dose was given over 30 minutes and the remaining 80% of the dose was given over the next 60 minutes, for a total infusion time of 90 minutes. Commercial preparations of rituximab were used.
Drug: CHOP (cyclophosphamide, hydroxydaunorubicin [doxorubicin], Oncovin [vincristine], prednisone) — Commercial preparations of CHOP were used. Prednisone was administered prior to rituximab infusion.
Drug: CVP (cyclophosphamide, vincristine, prednisone) — Commercial preparations of CVP were used. Prednisone was administered prior to rituximab infusion.
Drug: Analgesic/antipyretic and antihistamine drugs — An analgesic/antipyretic (eg, acetaminophen) and an antihistamine (eg, diphenhydramine) were administered 30 minutes before each infusion of rituximab.

SUMMARY:
This was a prospective, open-label, Phase III, multicenter, single-arm trial designed to assess the safety, pharmacokinetics, and pharmacodynamics of an alternative dosing rate of rituximab in previously untreated patients with diffuse large B-cell lymphoma (DLBCL) and follicular non-Hodgkin lymphoma (NHL).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥ 18 years
* Patients with previously untreated diffuse large B-cell lymphoma (DLBCL) who are scheduled to receive rituximab 375 mg/m^2 plus CHOP (cyclophosphamide, hydroxydaunorubicin [also called doxorubicin or adriamycin], Oncovin [vincristine], prednisone or prednisolone) chemotherapy, or previously untreated follicular non-Hodgkin lymphoma (NHL) who are scheduled to receive rituximab 375 mg/m^2 plus CVP (cyclophosphamide, vincristine, prednisolone) chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Clinically significant cardiovascular disease (eg, uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) Classification Grade II or greater congestive heart failure, a ventricular arrhythmia requiring medication within 1 year prior to Day 1, or NYHA Grade II or greater peripheral vascular disease on Day 1 (first day of treatment)

Patients who meet any of the following criteria will be excluded from further study participation after Cycle 1:

* Circulating lymphocyte count > 5,000/μL before the Cycle 2 rituximab infusion
* Development of a serious and/or Grade 3 or 4 adverse event during Cycle 1 judged by the investigator to be related to the rituximab infusion
* Prior premedication with additional corticosteroids other than the prednisone included in the chemotherapy regimens

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2008-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Hurst, M.D., Study Director — Genentech, Inc.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 451 enrolled patients, 26 withdrew before receiving treatment and are not included in the Baseline Characteristics nor any of the Outcome Measures.
Period: Enrolled in Study
Arm/Group | Rituximab 375 mg/m^2
Started | 451
Completed | 425
Not Completed | 26
Not completed — Physician decision to withdraw patient | 1
Not completed — Subject decision to withdraw | 8
Not completed — Various Reasons | 17
Period: Received Cycle 1 Treatment
Arm/Group | Rituximab 375 mg/m^2
Started | 425
Completed | 372
Not Completed | 53
Not completed — Adverse Event | 8
Not completed — Death | 5
Not completed — Eligibility criteria for Cycle 2 not met | 11
Not completed — Physician decision to withdraw patient | 7
Not completed — Subject decision to withdraw | 9
Not completed — Various Reasons | 13
Period: Received Cycle 2 Treatment
Arm/Group | Rituximab 375 mg/m^2
Started | 372
Completed | 304
Not Completed | 68
Not completed — Adverse Event | 12
Not completed — Death | 6
Not completed — Disease progression | 3
Not completed — Lost to Follow-up | 3
Not completed — Physician decision to withdraw patient | 13
Not completed — Subject decision to withdraw | 6
Not completed — Various Reasons | 25

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 425
Age, Continuous [Mean (Standard Deviation); unit: years] — Demographic data are reported for the intent-to-treat (ITT) population which included all patients who received at least 1 dose of rituximab regardless of infusion rate. Of the 451 enrolled patients, 26 withdrew before receiving treatment and were not included in the ITT population.
  years | 62.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic data are reported for the intent-to-treat (ITT) population which included all patients who received at least 1 dose of rituximab regardless of infusion rate. Of the 451 enrolled patients, 26 withdrew before receiving treatment and were not included in the ITT population.
  Participants
    Female | 191
    Male | 234

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Developed Grade 3 or 4 Infusion-related Reactions (IRR) Resulting From Faster Infusion of Rituximab During Days 1 and 2 of Cycle 2
Description: The percentage of patients who developed Grade 3 or 4 IRRs resulting from faster infusion of rituximab at Cycle 2 was assessed in patients who had previously received rituximab at the standard infusion rate without experiencing a Grade 3 or 4 IRR at Cycle 1. IRRs were a predefined list of Medical Dictionary for Regulatory Activities (MedDRA) terms for infusion-related adverse events occurring on the day of and/or the day after rituximab infusion. The list of IRR terms was compiled based on IRRs observed in the present and previous studies in which rituximab was infused at the standard rate.
Time Frame: Days 1 and 2 of Cycle 2
Population: Per-protocol evaluable population: All patients who received rituximab by faster infusion in Cycle 2 and who did not experience a Grade 3 or 4 infusion-related reaction during the rituximab infusion given at the standard rate during Cycle 1.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 363
Percentage of participants | 1.1 [0.3 to 2.8]

2. Secondary Outcome: Percentage of Patients Who Had an Adverse Event of Any Grade or Seriousness During Cycle 1
Time Frame: Cycle 1
Population: Intent-to-treat (ITT) population: All patients who received at least 1 dose of rituximab regardless of infusion rate.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 425
Percentage of participants | 91.8

3. Secondary Outcome: Percentage of Patients Who Had an Adverse Event of Any Grade or Seriousness During Cycle 2 Through Cycle 6 or 8 (End of Study)
Time Frame: Cycle 2 through Cycle 6 or 8 (end of study)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 363
Percentage of participants | 98.6

4. Secondary Outcome: Duration of Rituximab Infusion Including Dose Interruption Times
Description: The median duration of the rituximab infusion on Day 1 of each cycle, including the duration of dose interruptions, is reported.
Time Frame: Day 1 of each of Cycles 1 to 6 or 8
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 363
Minutes
  Cycle 1 (n=362) | 245 [225 to 273]
  Cycle 2 (n=363) | 91 [90 to 98]
  Cycle 3 (n=344) | 91 [90 to 98]
  Cycle 4 (n=329) | 91 [90 to 96]
  Cycle 5 (n=312) | 91 [90 to 95]
  Cycle 6 (n=303) | 91 [90 to 96]
  Cycle 7 (n=59) | 91 [90 to 95]
  Cycle 8 (n=59) | 91 [90 to 95]

5. Secondary Outcome: Maximum Serum Concentration (Cmax) of Rituximab Post-dose at the First Alternative Dosing Rate (Cycle 2) and the Last Cycle (Either Cycle 6 or 8)
Description: Serum samples for rituximab pharmacokinetic analysis were taken pre-dose (within 15 minutes before rituximab infusion) and post-dose (within 15 minutes after the end of the rituximab infusion) after the first faster infusion (Cycle 2) and after the last infusion (either Cycle 6 or 8). An enzyme-linked immunosorbent assay (ELISA) was used to measure rituximab levels in the serum samples.
Time Frame: Day 1 of Cycles 2 and either 6 or 8 (last cycle)
Population: Pharmacokinetic evaluable population: All patients who received at least 1 infusion of rituximab and had rituximab concentration data.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 335
µg/mL
  Cycle 2 (n=335) | 228.0 (63.7)
  Cycle 6 (n=238) | 275.0 (71.5)
  Cycle 8 (n=36) | 299.0 (90.6)

6. Secondary Outcome: Percentage of Patients Who Had Undetectable Levels of CD19+ Lymphocytes at Cycle 2 and Either Cycle 6 or 8 (Last Cycle)
Description: Serum samples for measurement of CD19+ lymphocytes were taken pre-dose (within 15 minutes before rituximab infusion). CD19+ lymphocyte counts were measured by flow cytometry using a fluorescent-activated cell sorter (FACS).
Time Frame: Day 1 of Cycle 2 and either Cycle 6 or 8 (last cycle)
Population: Per-protocol evaluable population: All patients who received rituximab by faster infusion in Cycle 2 and who did not experience a Grade 3 or 4 infusion-related reaction during the rituximab infusion given at the standard rate during Cycle 1. Only patients with pre-dose CD19+ lymphocyte counts at each time point were included in the analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab 375 mg/m^2
Number analyzed (Participants) | 338
Percentage of participants
  Cycle 2 (n=338) | 50.5 (24)
  Cycle 6 (n=240) | 68.3 (4)
  Cycle 8 (n=32) | 87.5 (0)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded from the start of study treatment until 30 days following the last administration of study treatment or at study discontinuation/early termination, whichever occurred earlier.
Description: Adverse events are reported for the intent-to-treat (ITT) population which included all patients who received at least 1 dose of rituximab, regardless of infusion rate.
Arm/Group | Rituximab 375 mg/m^2
Serious Adverse Events (participants affected / at risk) | 107/425
Other Adverse Events (participants affected / at risk) | 421/425
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=425)
Febrile neutropenia (Blood and lymphatic system disorders) | 33
Neutropenia (Blood and lymphatic system disorders) | 10
Pancytopenia (Blood and lymphatic system disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 2
Cardiac failure congestive (Cardiac disorders) | 3
Atrial fibrillation (Cardiac disorders) | 3
Cardiomyopathy (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Small intestinal obstruction (Gastrointestinal disorders) | 2
Pancreatitis (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal mass (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Small intestinal perforation (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Megacolon (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 3
Chest pain (General disorders) | 3
Asthenia (General disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 2
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Pneumonia (Infections and infestations) | 7
Bronchitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Device related sepsis (Infections and infestations) | 1
Fungal sepsis (Infections and infestations) | 1
Neutropenic sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Staphylococcal sepsis (Infections and infestations) | 1
Pseudomonal sepsis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 1
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 12
Failure to thrive (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 3
Jugular vein thrombosis (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1
Hypotension (Vascular disorders) | 2
Orthostatic hypotension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
Superior vena cava syndrome (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 375 mg/m^2 (N=425)
Neutropenia (Blood and lymphatic system disorders) | 135
Anaemia (Blood and lymphatic system disorders) | 100
Thrombocytopenia (Blood and lymphatic system disorders) | 55
Leukopenia (Blood and lymphatic system disorders) | 31
Nausea (Gastrointestinal disorders) | 202
Vomiting (Gastrointestinal disorders) | 69
Constipation (Gastrointestinal disorders) | 142
Diarrhoea (Gastrointestinal disorders) | 99
Abdominal pain (Gastrointestinal disorders) | 43
Dyspepsia (Gastrointestinal disorders) | 51
Stomatitis (Gastrointestinal disorders) | 34
Dry mouth (Gastrointestinal disorders) | 37
Fatigue (General disorders) | 227
Asthenia (General disorders) | 47
Pain (General disorders) | 30
Chest pain (General disorders) | 23
Pyrexia (General disorders) | 63
Chills (General disorders) | 49
Oedema peripheral (General disorders) | 44
Mucosal inflammation (General disorders) | 43
Upper respiratory tract infection (Infections and infestations) | 27
Candidiasis (Infections and infestations) | 22
Weight decreased (Investigations) | 33
Decreased appetite (Metabolism and nutrition disorders) | 72
Dehydration (Metabolism and nutrition disorders) | 36
Hypokalaemia (Metabolism and nutrition disorders) | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 26
Hyperglycaemia (Metabolism and nutrition disorders) | 23
Back pain (Musculoskeletal and connective tissue disorders) | 56
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24
Bone pain (Musculoskeletal and connective tissue disorders) | 41
Arthralgia (Musculoskeletal and connective tissue disorders) | 43
Muscle spasms (Musculoskeletal and connective tissue disorders) | 30
Neuropathy peripheral (Nervous system disorders) | 99
Peripheral sensory neuropathy (Nervous system disorders) | 37
Dysgeusia (Nervous system disorders) | 58
Headache (Nervous system disorders) | 75
Dizziness (Nervous system disorders) | 59
Paraesthesia (Nervous system disorders) | 33
Insomnia (Psychiatric disorders) | 100
Anxiety (Psychiatric disorders) | 42
Depression (Psychiatric disorders) | 22
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57
Cough (Respiratory, thoracic and mediastinal disorders) | 65
Alopecia (Skin and subcutaneous tissue disorders) | 169
Rash (Skin and subcutaneous tissue disorders) | 45
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 24
Pruritus (Skin and subcutaneous tissue disorders) | 28
Hypotension (Vascular disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.